CLINICAL TRIAL: NCT01028222
Title: The TEAM Trial (Tasigna Efficacy in Advanced Melanoma): A Phase II, Open Label, Multi-center, Single-arm Study to Assess the Efficacy of Tasigna ® in the Treatment of Patients With Metastatic and/or Inoperable Melanoma Harboring a c-Kit Mutation
Brief Title: A Study of AMNN107 in the Treatment of Metastatic and/or Inoperable Melanoma Harboring a c-Kit Mutation
Acronym: TEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAMN107B2301; 2009-015514-21 (EudraCT Number)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Melanoma
Keywords: Melanoma; AMN107; c-Kit; c-Kit mutated metastatic and/or inoperable melanoma
MeSH Terms: conditions — Melanoma | interventions — nilotinib; Dacarbazine

ARMS (2):
- Nilotinib (Experimental): 400 mg twice daily
  Interventions: Drug: Nilotinib
- DTIC (Active Comparator): 850 mg/m2 IV every 3 weeks
  Interventions: Drug: DTIC

INTERVENTIONS:
Drug: Nilotinib — Nilotinib was provided as 200 mg hard gelatin capsules for oral use.
  Other Names: AMN107
  Arms: Nilotinib
Drug: DTIC — DTIC was supplied locally as sterile powder for i.v. infusion.
  Other Names: Dacarbazine
  Arms: DTIC

SUMMARY:
The purpose of this study is to determine whether nilotinib is efficacious in the treatment of metastatic and/or inoperable melanoma harboring a c-Kit mutation.

DETAILED DESCRIPTION:
This trial began as a multi-center, randomized, Phase III, controlled trial for nilotinib vs (DTIC) dacarbazine to assess the efficacy and safety of nilotinib (400 mg bid) in patients with c-Kit mutated metastatic and/or inoperable melanoma. The study was open to patients with mucosal or acral melanoma.

Due to substantial difficulties identifying and recruiting eligible patients, the trial design was altered from a randomized, two-arm, Phase III study to a single-arm, Simon two-stage Phase II study with protocol Amendment 2 (27-Jul-2011). While the original protocol required the recruitment of 120 patients, this amendment required the study to recruit only 41 patients (patients randomized to nilotinib prior to Amendment 2 were to be counted in this total, but those randomized to dacarbazine ( DTIC ) DTIC were not). Patients randomized to DTIC were allowed to cross-over to nilotinib, either immediately or at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed mucosal or acral 2. Presence of a c-Kit mutation of exon 9, 11 or 13, or mutations Y822D and mutations D820Y, Y823D of exon 17, as confirmed by the central laboratory 3. Stage III unresectable or stage IV disease 4. The presence of one or more measurable lesions as detected by radiological or photographic methods and assessed according to RECIST 1.0. Lesions must have a size of at least 10mm at longest diameter (using a slice thickness of 5 mm)or double the slice thickness to be considered a target lesion. Target lesions should not be selected in previously irradiated fields unless there is clear evidence of progression 5. WHO performance status 0 - 2

Exclusion Criteria:

1. C-Kit mutation of exons 17(except mutations D820Y, Y822D or Y823D) or any other exon not allowed by the inclusion criteria
2. Patients with c-Kit amplifications only and no mutation
3. Patients with any history of brain metastases
4. Patients who have had any prior treatment with TKIs
5. Patients receiving medications or herbal extracts which interfere with nilotinib metabolism which are not discontinued by the time of the baseline visit
6. Acute or chronic liver or renal disease considered unrelated to melanoma

Other protocol-defined inclusion/exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (14):
  - City of Hope National Medical Center City of Hope national Med Ctr, Duarte, California
  - University of California San Diego - Moores Cancer Center UCSD Moores Cancer Center, La Jolla, California
  - University of California at Los Angeles UCLA, Los Angeles, California
  - California Pacific Medical Center California Pacific Med, San Francisco, California
  - University of Colorado Univ Colorado 2, Aurora, Colorado
  - Rush University Medical Center SC, Chicago, Illinois
  - Oncology Specialists, SC Dept.of Oncology Specialists, Park Ridge, Illinois
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. Medical Oncology, Baltimore, Maryland
  - Dana Farber Cancer Institute DFCI - Brookline, Boston, Massachusetts
  - Mayo Clinic - Rochester Mayo Clinic- Gonda, Rochester, Minnesota
  - Washington University School of Medicine CAMN107B2301, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve Case Western, Cleveland, Ohio
  - Baylor Health Care System/Sammons Cancer Center Baylor 2, Dallas, Texas
- Novartis Investigative Site, Buenos Aires, Buenos Aires, Argentina
- Australia (4):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Beijing, China
- Germany (5):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- Italy (5):
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Siena, SI
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- [Derived] Guo J, Carvajal RD, Dummer R, Hauschild A, Daud A, Bastian BC, Markovic SN, Queirolo P, Arance A, Berking C, Camargo V, Herchenhorn D, Petrella TM, Schadendorf D, Sharfman W, Testori A, Novick S, Hertle S, Nourry C, Chen Q, Hodi FS. Efficacy and safety of nilotinib in patients with KIT-mutated metastatic or inoperable melanoma: final results from the global, single-arm, phase II TEAM trial. Ann Oncol. 2017 Jun 1;28(6):1380-1387. doi: 10.1093/annonc/mdx079. PMID 28327988
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib | DTIC
Started | 42 | 13
Cross Over From DTIC to Nilotinib | 0 | 10
Completed | 4 | 0
Not Completed | 38 | 13
Not completed — Protocol deviation | 1 | 0
Not completed — Disease progression | 33 | 9
Not completed — Administrative problems | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Crossover to nilotinib w/out progression | 0 | 2
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | DTIC | Total
Number analyzed (Participants) | 42 | 13 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (12.39) | 68.8 (12.99) | 66.8 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 19 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the proportion of participants with a best overall response (BOR) of a confirmed complete response or partial response (CR+PR) determined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) based on local investigators' assessment (CT/MRI/photography). Per RECIST, CR: disappearance of all target lesions, all non-target lesions, and no new lesion; PR: a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no unequivocal progression of non-TLs, and no new lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments at least 4 weeks apart.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Participants
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Participants | 11 | 3

2. Secondary Outcome: Durable Overall Response Rate (DORR)
Description: DORR was defined as the rate of best overall response (CR+PR) lasting at least 12 weeks determined by RECIST v1.0 based on local investigators' assessment (CT/MRI/photography). The duration of ORR responders is computed from the date of first documented response (CR/PR) to the date of first documented progression or death due to underlying disease. Per RECIST, CR: disappearance of all target lesions, all non-target lesions, and no new lesion; PR: a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no worsening of non-TLs, and no new lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments at least 4 weeks apart.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Participants
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Participants | 11 | 3

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. Progression is defined using RECIST v1.0, as a >=20% increase in the sum of longest diameter of all target lesions, from smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or unequivocal progression of non-target lesions.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Months | 4.2 [2.1 to 5.8] | 4.2 [0.8 to 8.0]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the start of treatment to the date of death due to any cause.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Months | 18.0 [10.9 to 20.3] | 22.8 [4.9 to NA] — The 95% Confidence upper interval could not be calculated because there were too few events.

5. Secondary Outcome: Time to Objective Response (TOR)
Description: TOR was defined as the time between the start date of treatment until first documented confirmed response of CR or PR determined by RECIST v1.0 based on local investigators' assessment (CT/MRI/photography). Per RECIST, CR: disappearance of all target lesions, all non-target lesions, and no new lesion; PR: a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no unequivocal progression of non-TLs, and no new lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments at least 4 weeks apart.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
months | NA [NA to NA] — The TOR median could not be reached because there were too few events. | NA [NA to NA] — The TOR median could not be reached because there were too few events.

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with an overall response of CR of any duration, PR of any duration, or stable disease (SD) for a minimum of 12 weeks from start of treatment. Per RECIST, CR: disappearance of all target lesions, all non-target lesions, and no new lesion; PR: a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no unequivocal progression of non-TLs, and no new lesions; PD, a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; SD: no change or small changes that do not meet previously given criteria for CR, PR or PD.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Participants
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Participants | 20 | 7

7. Secondary Outcome: PFS Rate
Description: as for outcome 3
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Percentage of participants | 34.6 | 23.1

8. Secondary Outcome: OS Rate
Description: OS was defined as the time from the date of the start of treatment to the date of death due to any cause.
Time Frame: End of study (up to 39 months)
Population: Full analysis set (FAS): The FAS included all participants to whom treatment was assigned.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib | DTIC
Number analyzed (Participants) | 42 | 13
Percentage of participants | 63.6 | 66.7

ADVERSE EVENTS:
Groups:
- Crossover Nilotinib Treatment: Crossover nilotinib treatment
Arm/Group | Nilotinib | DTIC | Crossover Nilotinib Treatment
Serious Adverse Events (participants affected / at risk) | 12/42 | 1/13 | 4/10
Other Adverse Events (participants affected / at risk) | 40/42 | 9/13 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=42) | DTIC (N=13) | Crossover Nilotinib Treatment (N=10)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=42) | DTIC (N=13) | Crossover Nilotinib Treatment (N=10)
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 18 | 5 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 1 | 1
Asthenia (General disorders) | 2 | 1 | 3
Chills (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 13 | 5 | 4
Feeling cold (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 2
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 3 | 2
Suprapubic pain (General disorders) | 1 | 0 | 1
Temperature intolerance (General disorders) | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2
Oral fungal infection (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 10 | 1 | 1
Amylase increased (Investigations) | 8 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 1 | 0
Bilirubin conjugated increased (Investigations) | 11 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 0 | 0
Blood bilirubin increased (Investigations) | 19 | 1 | 3
Blood bilirubin unconjugated increased (Investigations) | 9 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 4 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 4 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 11 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 2
Lipase increased (Investigations) | 8 | 1 | 2
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Total bile acids increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 5 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 20 | 2 | 3
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 0 | 2
Lymphoedema (Vascular disorders) | 1 | 1 | 0
Vein disorder (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.